CLINICAL TRIAL: NCT05806463
Title: Efficacy of a Simplified Cognitive Behavioral Therapy Approach to Support Postpartum Mental Health and Address Social and Behavioral Barriers to Postpartum Family Planning in Ethiopia: A Cluster Randomized Controlled Trial
Brief Title: Efficacy of Mother's Time in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Johns Hopkins Center for Communication Programs (Unknown); Camber Collective (Other); DeepDive Consulting (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23020
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Depression, Postpartum; Anxiety, Postpartum; Contraceptive Usage
Keywords: Postpartum depression; Postpartum anxiety; Postpartum family planning
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders; Contraception Behavior

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized parallel intervention study model.
  Following random assignment of clusters to either the intervention or control arm and subsequent recruitment of participants, individuals will be enrolled in the study.
  Intervention arm: Mother's Time intervention Control arm: Standard of care
  Clusters will be randomly assigned using a random number generator to either the intervention arm or the control arm. Then, all individuals recruited within a given cluster will be assigned to the same intervention condition.
  Anticipating that the Mother's Time intervention will be superior to the standard care with respect to reducing symptoms of stress, depression, and anxiety and increasing modern contraceptive use, women in the control group will have opportunity to receive the full intervention upon completion of the intervention to the intervention group.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be fully blinded to whether participants are in an intervention or control cluster. However, the use of a cluster-randomized approach reduces the risk of contamination among women from different clusters because it reduces the risk of communication between individuals in intervention and control arms. As HEWs will be responsible for assisting with recruitment of participants, HEWs will be aware of these eligibility criteria and who has been recruited for the study in both the control and intervention arms. As a result, HEWs will not be fully blinded to the study. Outcome assessors and statisticians will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother's Time Intervention (Experimental): Working with local research partners, the research team will train HEWs in the intervention clusters in the Amhara region of Ethiopia to deliver four intervention sessions in a group setting of approximately six to eight women (average: 7). These sessions will take place over a period of approximately one month. Participants in the intervention group will receive four sessions of Mother's Time, delivered by an HEW.
  Interventions: Behavioral: Mother's Time
- Standard of care (No Intervention): Participants in the control group will receive the standard of care that postpartum mothers in Ethiopia receive. Standard of care for postpartum mothers related to family planning and mental health in Ethiopia includes multiple touch points that correspond with postpartum care as well as routine immunization.

INTERVENTIONS:
Behavioral: Mother's Time — Mother's Time is an evidence-based cognitive behavioral therapy (CBT) tool designed to support postpartum women experiencing mild to moderate symptoms of stress, depression, or anxiety. The intervention is designed for use by Ethiopian community health workers (CHWs) and includes CBT exercises and discussion on topics relating to family planning, such as planning for the future, speaking to the husband, and considering potential side effects.
  Arms: Mother's Time Intervention

SUMMARY:
Mother's Time is an evidence-based cognitive behavioral therapy (CBT) tool designed to support postpartum women experiencing mild to moderate symptoms of stress, depression or anxiety. The intervention is designed for use by Ethiopian community health workers (CHWs) and includes CBT exercises and discussion on topics relating to family planning, such as planning for the future, speaking to the husband, and considering potential side effects.

The primary objective of this research is to test the efficacy of Mother's Time, on mild to moderate symptoms of postpartum stress, anxiety, and depression as well as associated behavioral and social barriers to postpartum family planning, specifically among women under 25 who have given birth within the last year.

DETAILED DESCRIPTION:
Mother's Time is an evidence-based cognitive behavioral therapy (CBT) tool designed to support postpartum women experiencing mild to moderate symptoms of stress, depression, or anxiety. The intervention is designed for use by Ethiopian community health workers (CHWs) and includes CBT exercises and discussion on topics relating to family planning, such as planning for the future, speaking to the husband, and considering potential side effects.

The primary objective of this research is to test the efficacy of Mother's Time, on mild to moderate symptoms of postpartum stress, anxiety, and depression as well as associated behavioral and social barriers to postpartum family planning, specifically among women under 25 who have given birth within the last year. This study builds on evidence from a previous study (Principal Investigator: Hendrickson, Institutional Review Board (IRB) #: 16604) demonstrating the feasibility and acceptability of using Mother's Time to address mild to moderate depressive and anxiety symptoms and associated behavioral and social barriers to family planning in Ethiopia. The study also builds on previous human-centered design work (Principal Investigator: Hendrickson, IRB #: 21414) to obtain further design input on the Mother's Time intervention. The investigators have adapted the intervention based on data and findings from the pilot study and the Human Centered Design workshop. The specific aims of this study are to:

1) Quantitatively examine the impact of participating in Mother's Time on symptoms of stress, depression, and anxiety among postpartum women ages 16-24 years of age who have given birth within the last year.

1a) Assess the immediate (post intervention) and longer term (3-month post-intervention) impact of participation in Mother's Time on symptoms of stress, depression, and anxiety.

2) Quantitatively assess the impact of participating in Mother's Time on use of a modern contraceptive method among postpartum women ages 16-24 years of age who have given birth within the last year.

2a) Assess the immediate (post intervention) and longer term (3-month post-intervention) impact of participation in Mother's Time on use of a modern contraceptive method among postpartum women.

2b) Quantitatively assess the impact of participating in Mother's Time on perceived benefits and self-efficacy to engage in healthy thinking patterns and modify behaviors related to family planning.

3) Explore feasibility and acceptability of implementing Mothers Time from the perspective of health extension workers (HEWs) and HEW supervisors.

ELIGIBILITY:
Inclusion Criteria:

* Has given birth within the last year to an infant who is still living
* Not currently using a method of modern family planning (Women who are breastfeeding but not following the Lactation Amenorrhea Method (LAM) criteria will be considered "not using")
* Married (traditional, religious or legal)
* Aged 16-24 (participants under 18 will be considered emancipated minors as these individuals will be married)
* Scores between 5 and 14 on the PHQ-9 questionnaire and/or between 5 and 14 on the GAD-7 questionnaire
* In screener, does not indicate she has "death ideation" ("no" response on question 14) Consents to participate in study

Exclusion Criteria:

* Unmarried women
* Women under age 16 or over age 24
* Women who have lost their infants since birth
* Scores under 5 on both the PHQ-9 and GAD-7 questionnaire
* Scores over 14 on both the PHQ-9 and GAD-7 questionnaire
* In screener, indicates she has "death ideation" ("yes" response on question 14)

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 328 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in postpartum depression | Baseline, Endline up to 1 month post-intervention, 3-month follow-up
  Symptoms of depression using Patient Health Questionnaire-9 (PHQ-9). This is a 9-item questionnaire with scores for each question ranging from 0 (not at all) to 3 (nearly every day). Scores are summed for an overall score range of 0-27, with higher scores meaning more greater depression severity.
Change in postpartum anxiety | Baseline, Endline up to 1 month post-intervention, 3-month follow-up
  Symptoms of anxiety using General Anxiety Disorder-7 (GAD-7). This is a 7-item questionnaire with scores for each question ranging from 0 (not at all) to 3 (nearly every day). Scores are summed for an overall score range of 0-21, with higher scores meaning more greater anxiety severity.
Change in postpartum family planning | Baseline, Endline up to 1 month post-intervention, 3-month follow-up
  Current use of modern contraception method postpartum (yes vs. no)

CONTACTS AND LOCATIONS:
Overall Officials: Stella Babalola, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Health centers/clusters in selected woredas, West Gojjam, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No
The investigators plan to share summary reports and presentations about this research project and results in presentations to the investigators' funder, USAID, local partners, the Ethiopian Ministry of Health and other stakeholders working in family planning, mental health, or maternal health. All shared information will be at the summary level and not provide any identifiable information. The investigators also plan to publish peer-reviewed articles and international comments which will not include any identifiable information. If journal reviewers request data, the investigators will provide high-level, aggregated descriptive statistics on our participants from the quantitative data, but will not share full datasets or transcripts outside the study team. As these data are related to a potentially sensitive topic, they will not be made publicly available. Due to the relatively small sample size, making data publicly available could create risks around confidentiality.